CLINICAL TRIAL: NCT03917693
Title: A Human Intervention Trial Investigating the Effects of Phytin on the Human Gut Microbiome
Brief Title: Effect of Phytin on Human Gut Microbiome (EPoM)
Acronym: EPoM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: QIB03-2018
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Diet Modification
MeSH Terms: interventions — Phytic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This process will be carried out by a QIB scientist who is not part of the study team.
  Wendy Hollands (QIB Food Innovation and Health [FIH] scientist) will be responsible for this process, and therefore ensures the trial remains blinded to the study participants, Chief Investigators and study scientists/advisors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phytin capsules (Active Comparator): 2.4 g phytin to be consumed daily for a period of 2 weeks. Participants will consume 2 test capsules containing phytin, 3 times a day with a meal for a period of 2 weeks.
  Interventions: Dietary Supplement: Phytin, rice extract
- Microcrystalline cellulose (MCC) capsules (Placebo Comparator): 2.4 g MCC to be consumed daily for a period of 2 weeks. Participants will consume 2 placebo capsules, each containing microcrystalline cellulose, 3 times a day with a meal for a period of 2 weeks.
  Interventions: Other: MCC, placebo

INTERVENTIONS:
Dietary Supplement: Phytin, rice extract — Consumption of a rice extract, called phytin for a period of 2 weeks
  Arms: Phytin capsules
Other: MCC, placebo — Consumption of MCC, a placebo, for a period of 2 week
  Arms: Microcrystalline cellulose (MCC) capsules

SUMMARY:
Within many plants, such as seeds, nuts and cereals, there is a compound called phytic acid. Phytic acid has many beneficial properties, including producing molecules which slows down the damage that can be caused to other molecules within the body. Phytic acid has also been known to help in the treatment of cancer. Phytic acid binds iron very strongly. Iron is an extremely important nutrient not only for humans, but also for a lot of bacteria. In humans, iron is absorbed in the small intestine. Unfortunately, iron does not get absorbed very well and so a lot of it travels into the large intestine. The large intestine contains trillions of bacteria and a lot of these bacteria use iron as food. However, not all bacteria in the large intestine are 'good bacteria'. Some bacteria, such as Enterobacteria, can be harmful to people's health. For this reason, if iron is kept away from these 'bad bacteria' through the binding of phytic acid and iron, it could prove to be beneficial to human health. In general, the gut contains trillions of bacteria, many of which help to unlock extra nutrients from the food people eat. Some bacteria, such as Bifidobacteria, are often referred to as 'good bacteria' and are added to foods such as yoghurts. Many 'good bacteria' are able to survive without iron and this makes it even more important to make sure the 'bad bacteria' have limited access to iron. Otherwise, it is possible that the large intestine could populate more more harmful bacteria than beneficial bacteria.

In this study, investigators will ask participants to consume either the test capsule, which contains phytin (a salt form of phytic acid), or a control capsule, which contains a powder resembling phytin but is actually an inactive substance. The investigators are interested in whether consuming these capsules will decrease Enterobacteria (one of the 'bad bacteria' in the large intestine).

DETAILED DESCRIPTION:
The study will take place at the Clinical Research Facility (CRF) at the Quadram Institute in Norwich, with participants attending the QI CRF for screening and to collect the capsules for consumption (capsules will be randomly allocated, containing either phytin or placebo (microcrystalline cellulose)). The participants will be recruited from within a 40-mile radius of Norwich and this is clearly stated in the Participant Information Sheet (PIS). In this study, male and female participants aged between 18 and 50 years will be recruited until 14 participants complete the study. The participants will consume the randomly allocated capsules (containing either phytin or placebo), and collect their faecal samples at their home.

The purpose of this study is to ascertain whether the delivery of phytin to the colon will cause a decrease in the proportions of human gut enterobacteriaceae, and a potential concomitant increase in the proportion of human gut bifidobacteriaceae, through chelation of iron.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 50
* Non-smokers (e-cigarette/vape users are able to participate)
* Those with a body mass index (BMI) between 19.5 and 30 kg/m^2
* Those that live within a 40-mile radius of Norwich

Exclusion Criteria:

* results of our screening test indicate the participant is not suitable to take part in this study
* are pregnant, have been pregnant in the last year or are lactating and/or breast feeding
* are currently suffering from, or have ever suffered from, any diagnosed gastrointestinal disease, gastrointestinal disorders including regular diarrhoea and constipation (excluding hiatus hernia unless symptomatic), and/or have undergone gastrointestinal surgery, or the study intervention/procedure is contraindicated
* have been diagnosed with any long-term medical condition that may affect the study outcome (e.g. cancer, diabetes, haemophilia, cardiovascular disease, glaucoma, anaemia). These will be assessed on an individual basis
* have been diagnosed with any long-term medical condition requiring medication that may affect the study outcome
* regularly taking over the counter medications for digestive/gastrointestinal conditions
* are on long-term antibiotic therapy. Participant may be able to take part if 4 weeks has passed from the end of a course of antibiotics (this will be assessed on an individual basis)
* regularly take laxatives (once a month or more)
* take certain dietary supplements or herbal remedies and are unwilling to stop taking them for one month prior to and during study period. This will be assessed on an individual basis
* take pre- or pro-biotic drinks &/or yoghurts on an occasional basis, unless willing to abstain for one month prior to and during the study period. (if participant regularly takes pre-&/or pro biotics (3+ times a week, and for more than one month) and will continue throughout the study then participant will not be excluded)
* are on or plan to start a diet programme that may affect the study outcome (e.g. 5:2 fasting diet) unless willing to abstain for 1 month prior to and during study period. This will be assessed on an individual basis
* recently returned to the United Kingdom (UK) following a period abroad, and who have suffered gastric symptoms during the period abroad or on return to the UK. These will be assessed on an individual basis
* regular/recent (within 3 months) use of colonic irrigation or other bowel cleansing techniques
* are involved in another research project that includes dietary intervention or involving blood sampling
* record blood in participant's stools or have two or more episodes of constipation or diarrhoea (type 1, 2, or 7 stools) during the study
* are unwilling to provide their General Practioner's (GP's) contact details
* are unable to provide written informed consent.
* regularly consume more than 15 units (women) or 22 units (men) of alcohol a week
* Regularly taking iron supplements
* Those unable to swallow capsules
* Those with abnormal blood pressure measurements (160/100 will be regarded as an exclusion value)
* Are related to someone in the study (e.g. spouse, partner, immediate family member)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Relative abundance of Enterobacteriaceae | 4 months
  To investigate whether consuming phytin for two weeks will cause a proportional decrease in human gut Enterobacteriaceae compared to the number of Enterobacteriaceae present in the participants' gut microbiome after consuming the control capsule.

SECONDARY OUTCOMES:
Relative abundance of Bifidobacteriaceae | 4 months
  To investigate whether the delivery of phytin to the colon for a period of two weeks will be associated with an increase in human gut bifidobacteriaceae through the chelation of iron, compared to the number of bifidobacteriaceae present in the participants' baseline gut microbiota, as determined by faecal bacteria phylogenic analysis
Gut microbial composition | 4 months
  To ascertain whether consuming phytin modulates the gut microbial community as a whole, as compared to the consumption of a placebo capsule
Short chain fatty acids | 4 months
  To determine whether the consumption of phytin causes a change in short chain fatty acid levels in the faeces, via changes in the gut microbiome function
Iron concentrations | 4 months
  To determine whether the consumption of phytin causes a change in the available iron present in the faeces
Phytin degradation | 4 months
  To ascertain the extent of phytin degradation that takes place in the colon based on the known concentration of phytin administered via the capsule
Gut inflammation | 4 months
  To determine levels of calprotectin as a marker of gut inflammation
Systemic inflammation | 4 months
  To determine levels of C-Reactive Protein (CRP) as a marker of systemic inflammation
Release of capsule | 4 months
  To measure serum ferritin levels as a marker of the time of capsule release

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Narbad, Prof, Study Chair — Quadram Institute Bioscience; Melanie Pascale, PhD, Principal Investigator — Quadram Institute Clinical Research Facility
Locations (2):
- United Kingdom (2):
  - Quadram Institute Bioscience, Norwich, Norfolk
  - QI NNUHFT Clinical Research Facility, Norwich, Norfolk